CLINICAL TRIAL: NCT00847184
Title: Comparison of Airtraq vs. MacIntosh Intubation Via Nasal Approach
Brief Title: Comparison of Airtraq Versus MacIntosh Intubation Via Nasal Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Prof. Dr. Harald Groeben, Kliniken Essen-Mitte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Airtraqnasal2009
Record Dates: First submitted 2009-02-11; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Tracheal Intubation
Keywords: nasal intubation; Aitraq; difficult intubation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Airtraq (Active Comparator): Intubation with the use of the Airtraq technique
  Interventions: Device: Airtraq
- 2. MacIntosh (Active Comparator): Intubation using the standard MacIntosh blade
  Interventions: Device: Intubation

INTERVENTIONS:
Device: Intubation — Intubation using the standard MacIntosh blade
  Arms: 2. MacIntosh
Device: Airtraq — Intubation with the use of the Airtraq technique
  Other Names: Aitraq, Prodol Meditec S.A., Vizcaya, Spain
  Arms: 1. Airtraq

SUMMARY:
Time, success rate, and number of optimising maneuvers for tracheal intubation via the nasal approach are not different when Aitraq technique is used compared to a standard MacIntosh blade.

DETAILED DESCRIPTION:
One hundred adult patients with an expected easy intubation and 100 patients with an expected difficult intubation are enrolled. Intubations are performed by two experienced fully boarded anesthesiologists. The design of the study is prospective and randomised.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for nasal intubation
* Adult

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Time for intubation | 10 month

SECONDARY OUTCOMES:
Success rate for intubation | 10 month

CONTACTS AND LOCATIONS:
Overall Officials: Harald Groeben, M.D., Principal Investigator — Kliniken Essen-Mitte
Locations (1):
- Prof. Dr. Harald Groeben, Essen, Germany

REFERENCES:
- [Background] Maharaj CH, Higgins BD, Harte BH, Laffey JG. Evaluation of intubation using the Airtraq or Macintosh laryngoscope by anaesthetists in easy and simulated difficult laryngoscopy--a manikin study. Anaesthesia. 2006 May;61(5):469-77. doi: 10.1111/j.1365-2044.2006.04547.x. PMID 16674623